CLINICAL TRIAL: NCT01544543
Title: Validation of HealthCare Standards in COPD
Brief Title: Validation of HealthCare Standards in Chronic Obstructive Pulmonary Disease
Acronym: VESALIO
Status: Completed | Type: Observational
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Juan José Soler Cataluna, MD, PhD, Sociedad Española de Neumología y Cirugía Torácica
Other Study IDs: VES0109
Record Dates: First submitted 2012-02-21; First posted 2012-03-06 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD Exacerbation Cohort: Patients hospitalized for a COPD exacerbation

SUMMARY:
VESALIO is a pilot study aimed at evaluating the feasibility and reliability (time stability and interobserver reliability) of healthcare quality standards in chronic obstructive pulmonary disease (COPD) recently outlined by SEPAR (Spanish Pneumology and Thoracic Surgery Society), and at establishing the foundation for a future validation (construct and criterion validation) of the aforementioned standards.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 40 years of age or older
* Diagnosis of COPD at hospital discharge
* Hospitalization for a COPD exacerbation

Exclusion Criteria:

* Patients hospitalized for the first time at the participating site without a documented history of COPD
* Patients currently participating of having ever participated in a COPD-related clinical trial
* Patients with a serious disease that might affect the measured outcomes (terminal oncologic disease, neoplastic disease for which the patient is receiving chemo/radiotherapy, terminal renal insufficiency, AIDS)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients hospitalized for an exacerbation of COPD
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2010-02

PRIMARY OUTCOMES:
COPD exacerbation | Within 12 months after hospitalization
Mortality | within 90 and 180 days after hospitalization
Healthcare-associated cost | within 12 months after hospitalization
  Hospital-stay lenght ER visits

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Soler Cataluna, MD, PhD, Principal Investigator — Hospital de Requena, Valencia
Locations (1):
- Hospital General de Requena, Requena, Valencia, Spain